CLINICAL TRIAL: NCT05088577
Title: Evaluation of the Effects of Egg Consumption and Its Enrichment With Annatto on Biomarkers of Cardiovascular Risk and Satiety in Adults.
Brief Title: Evaluation of Egg Consumption and Its Enrichment With Annatto on Cardiovascular Risk and Satiety in Healthy Adults
Acronym: EGGANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Principal Investigator, Jacqueline Barona Acevedo, Principal Investigator, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 754-2018; 111580763245 (Other Grant/Funding Number: Minciencias)
Record Dates: First submitted 2021-08-30; First posted 2021-10-22 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers
Keywords: Egg; Bixa orellana; Annatto; cardiovascular risk factors; clinical trial

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole egg (Experimental): Two whole eggs (50g each) to be eaten daily during 8 weeks
  Interventions: Dietary Supplement: Whole egg
- Annatto-enriched egg (Experimental): Two whole eggs (50g each) enriched with annatto (Bixa orellana L.) to be eaten daily during 8 weeks. Dose of annatto: 1,2 mg bixin/kg of body weight.
  Interventions: Dietary Supplement: Annatto-enriched egg
- Egg whites - Control (Placebo Comparator): Two egg whites to be eaten daily during 8 weeks
  Interventions: Dietary Supplement: Egg whites - Control

INTERVENTIONS:
Dietary Supplement: Whole egg — Daily consumption of two whole eggs during 8 weeks
  Arms: Whole egg
Dietary Supplement: Annatto-enriched egg — Daily consumption of two whole eggs enriched with annatto during 8 weeks
  Arms: Annatto-enriched egg
Dietary Supplement: Egg whites - Control — Daily consumption of two eggs whites during 8 weeks
  Arms: Egg whites - Control

SUMMARY:
Healthy adult volunteers (n= 105; 18-59 years) were randomly allocated to consume daily for 8 weeks, either two whole eggs (egg group), two whole eggs added with annatto (annatto-enriched egg group), or two egg whites (control). Volunteers were asked to continue with the habitual physical activity and diet, except for the consumption of additional eggs, egg whites or annatto.

It is hypothesized that participants consuming eggs would have a less atherogenic lipid profile, feel more satisfied and increase antioxidant levels in blood, compared to the control group. Participants in the annatto-enriched egg group would have greater antioxidant capacity than the egg group and compared to control.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-59 years
* Body Mass Index (BMI): 18,5 - 29,9 kg/m2
* Healthy volunteers
* Good disposition to consume either eggs, egg whites or eggs added with annatto
* To have signed the informed consent

Exclusion Criteria:

* Fasting blood triglycerides > 500mg/dL, Total Cholesterol > 240mg/dL, glucose > 126mg/dL or diabetes.
* Blood pressure: >140/90 mmHg.
* History or having any of the following: liver, kidney, or heart disease, cancer, endocrine or gastrointestinal disorders -especially those that limit food absorption.
* Use of medications to lower blood lipids or glucose.
* Consumption of multivitamins or nutraceuticals.
* Plan to lose body weight, pregnancy or breastfeeding.
* Any known allergy or intolerance to eggs or annatto.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Total cholesterol | Change from Baseline Total cholesterol at 8 weeks
  Fasting blood total cholesterol in mg/dL
Low-density lipoprotein (LDL) cholesterol | Change from Baseline LDL cholesterol at 8 weeks
  Fasting blood LDL cholesterol in mg/dL
Very low-density lipoprotein (VLDL) cholesterol | Change from Baseline VLDL cholesterol at 8 weeks
  Fasting blood VLDL cholesterol in mg/dL
Triglycerides | Change from Baseline Triglycerides at 8 weeks
  Fasting blood triglycerides in mg/dL
High-density lipoprotein (HLDL) cholesterol | Change from Baseline HDL cholesterol at 8 weeks
  Fasting blood HLDL cholesterol in mg/dL
Glucose | Change from Baseline Glucose at 8 weeks
  Fasting blood glucose in mg/dL
Systolic Blood Pressure | Change from Baseline Systolic Blood Pressure at 8 weeks
  Systolic blood pressure in mmHg will be used to present the results of this variable, as follow: e.g. 130 mmHg
Diastolic Blood Pressure | Change from Baseline Diastolic Blood Pressure at 8 weeks
  Diastolic blood pressure in mmHg will be used to present the results of this variable, as follow: e.g. 85 mmHg
Body Mass Index (BMI) in kg/m^2: weight in kilograms, height in meters | Change from Baseline BMI at 8 weeks
  weight and height will be combined to report BMI in kg/m^2
Waist circumference | Change from Baseline Waist circumference at 8 weeks
  Waist circumference in centimeters measured at the superior border of the iliac crest
Blood lutein levels | Change from Baseline Blood lutein levels at 8 weeks
  Fasting blood lutein levels in micrograms per mL
Dietary lutein+zeaxanthin levels | Change from Baseline Dietary lutein+zeaxanthin levels at 8 weeks
  Dietary lutein+zeaxanthin levels in micrograms
Blood bixin levels | Change from Baseline Blood bixin levels at 8 weeks
  Fasting blood bixin levels in %
Triglyceride-Rich lipoprotein (TRLP) size | Change from Baseline TRLP size at 8 weeks
  Fasting blood subclasses (Large, medium, small) of TRLP in nmol/L measured by Nuclear Magnetic Resonance
Low-density lipoprotein (LDL) size | Change from Baseline LDL size at 8 weeks
  Fasting blood subclasses (Large, medium, small) of LDL in nmol/L measured by Nuclear Magnetic Resonance
High-density lipoprotein (HDL) size | Change from Baseline HDL size at 8 weeks
  Fasting blood subclasses (Large, medium, small) of HDL in μmol/L measured by Nuclear Magnetic Resonance
Apolipoprotein B (ApoB) | Change from Baseline ApoB at 8 weeks
  Fasting blood ApoB in mg/L measured by Nuclear Magnetic Resonance
Apolipoprotein A1 (ApoA1) | Change from Baseline ApoA1 at 8 weeks
  Fasting blood ApoA1 in mg/L measured by Nuclear Magnetic Resonance
Ghrelin | Change from Baseline Ghrelin at 8 weeks
  Ghrelin in pg/mL
Visual Analog Scale (VAS) to Measure Perceived Hunger and Satiety | Change from Baseline VAS of Hunger and Satiety at 8 weeks
  "Visual Analog Scale to measure perceived hunger and satiety" to complete in the morning, fasting, 5 days before entering the study and the last 5 days to end the study (8th week). The VAS consist of 8 questions followed each by a line of 10cm in which the person marks a position corresponding to his/her feelings about hunger and satiety. A higher score (10) means the person feels with more hunger or satisfied.

SECONDARY OUTCOMES:
Ancestry Informative Marker | Baseline
  Percentage of genetic ethnicity of European, Amerindian and African for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Barona-Acevedo, PhD, Principal Investigator — Universidad de Antioquia
Locations (1):
- Sede de Investigación Universitaria - Universidad de Antioquia, Medellín, Antioquia, Colombia